CLINICAL TRIAL: NCT03963544
Title: Patterns of Care and Outcomes of Patients With METAstatic Gastrointestinal Stromal Tumors (GIST) in a Real-life Setting: the METAGIST Observational Study
Brief Title: Patterns of Care and Outcomes of Patients With METAstatic Gastrointestinal Stromal Tumors (METAGIST)
Acronym: METAGIST
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: French Sarcoma Group (Other)
Responsible Party: Sponsor
Other Study IDs: IB2019-METAGIST
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Gastro Intestinal Stromal Tumor
MeSH Terms: interventions — Tyrosine Kinase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: oral tyrosine-kinase inhibitors (TKI) of KIT and PDGFR as per recommendations — oral tyrosine-kinase inhibitors (TKI) of KIT and PDGFR

SUMMARY:
Gastro intestinal stromal tumors (GIST) are rare mesenchymal tumors of the gastrointestinal tract characterized by somatic mutations in the gene encoding the KIT or the PDGFR alpha protein1. Treatment of localized forms relies on adequate surgery without tumor spillage and systemic treatment with imatinib according to risk of relapse defined by localization, tumor size and mitotic count, as well as mutational status. Advanced and relapsing forms are currently treated with oral tyrosine-kinase inhibitors (TKI) of KIT and PDGFR such as Imatinib, Sunitinib and Regorafenib. Over two decades significant changes in drug discovery have impacted treatment strategies, notably via patient's access to various clinical trials. The use of focal treatments such as surgery or interventional radiology with mini invasive procedure of oligometastasis is also being proposed in some cases.

There is no precise data on patterns of sequential treatments used, especially proportions of patients with metastatic GIST eventually benefiting from access to a clinical trial or a focal treatment strategy in the course of their disease, and their results in terms of survival on a real life national level.

Using the French sarcoma Group national database we aim at describing treatments strategies proposed patients with metastatic GIST in the real life setting.

Objectives include : (i) Description of clinico-biological profiles, patterns of care and modalities of treatment of patients with metastatic GIST in a real-life national setting and (ii) evaluation of patients outcome in terms of time to next treatment (TNT) and survival

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years old
* with a diagnosis of metastatic Gastrointestinal Stromal Tumor (metastatic at diagnostic or metastatic relapse)
* From 1990 to 2018

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: metastatic Gastrointestinal Stromal Tumor
Sampling Method: Non-Probability Sample
Enrollment: 492 (Actual)
Dates: Start 1990-01 (Actual); Primary Completion 2024-09 (Actual); Study Completion 2024-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maud Toulmonde, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Comprehensive Cancer Center, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Toulmonde M, Dinart D, Brahmi M, Verret B, Jean-Denis M, Ducimetiere F, Desolneux G, Meeus P, Palussiere J, Buy X, Bouhamama A, Gillon P, Dufresne A, Henon C, Le Loarer F, Karanian M, Ngo C, Mathoulin-Pelissier S, Bellera C, Le Cesne A, Blay JY, Italiano A. Evolution of Patterns of Care and Outcomes in the Real-Life Setting for Patients with Metastatic GIST Treated in Three French Expert Centers over Three Decades. Cancers (Basel). 2023 Aug 28;15(17):4306. doi: 10.3390/cancers15174306. PMID 37686582

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Metastatic Gastrointestinal Stromal Tumors (GIST): Participants with metastatic Gastrointestinal stromal tumors (GIST) treated in one of the three national coordinating centers from NETSARC (Institut Bergonié, Centre Léon Berard and Institut Gustave Roussy) from 1990 to 2018.
Period: Overall Study
Arm/Group | Participants With Metastatic Gastrointestinal Stromal Tumors (GIST)
Started | 492
Completed | 492
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Metastatic Gastrointestinal Stromal Tumors (GIST)
Number analyzed (Participants) | 492
Age, Continuous [Median (Full Range); unit: years] | 59 [19 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200
  Male | 292
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 492

OUTCOME MEASURES:

1. Primary Outcome: Time to Next Treatment (TNT)
Description: time from the systemic treatment onset to the next treatment or death due to any cause, whichever came first.
Time Frame: 10 years
Population: Participants who received systemic treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Metastatic Gastrointestinal Stromal Tumors (GIST)
Number analyzed (Participants) | 461
months | 26.7 [23.4 to 32.3]

2. Primary Outcome: Overall Survival (OS) Time
Description: the interval between the diagnosis of metastatic disease or the first-line systemic therapy onset and the time of death.
Time Frame: 10 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Metastatic Gastrointestinal Stromal Tumors (GIST)
Number analyzed (Participants) | 492
months | 83.4 [72.7 to 97.9]

3. Secondary Outcome: Treatment With a Systemic Therapy
Description: Proportion of metastatic patients treated with a systemic therapy
Time Frame: At diagnosis of metastatic disease
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Gastrointestinal Stromal Tumors (GIST)
Number analyzed (Participants) | 492
Participants | 461

4. Secondary Outcome: Proportion of Participants Included in a Clinical Trial
Description: Proportion of participants included in a clinical trial (other than the present study) during the course of their metastatic disease
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Metastatic Gastrointestinal Stromal Tumors (GIST)
Number analyzed (Participants) | 492
Participants | 269

ADVERSE EVENTS:
Time Frame: 10 years Adverse events (serious and non-serious) were not collected
Description: Adverse events (serious and non-serious) were not collected
Arm/Group | Participants With Metastatic Gastrointestinal Stromal Tumors (GIST)
All-Cause Mortality (participants affected / at risk) | 221/492
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03963544/Prot_SAP_000.pdf